CLINICAL TRIAL: NCT01218256
Title: Combined Resistance and Endurance Training in Patients With Type 2 Diabetes: A Pilot-study to Assess the Effects of 2 Different Resistance Protocols on Muscle Mass, Strength and Glycemic Control.
Brief Title: Secondary Prevention in Type 2 Diabetes: Comparison of Two Different Resistance Exercise Training Protocols
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Professor Josef Niebauer, MD, PhD, MBA, Institute of Sports Medicine, Prevention and Rehabilitation, Paracelsus Medical University, Lindhofstrasse 20, 5020 Salzburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UISM-2-2010
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2007-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes mellitus; type 2 diabetes; T2DM; resistance training; hypertrophy training; endurance training
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypertrophy resistance training (Active Comparator): Aerobic endurance training combined with hypertrophy resistance training in type 2 diabetes mellitus.
  Interventions: Other: Physical exercise training
- Endurance resistance training (Active Comparator): Aerobic endurance training combined with hypertrophy resistance training in type 2 diabetes mellitus.
  Interventions: Other: Physical exercise training

INTERVENTIONS:
Other: Physical exercise training — aerobic endurance training (cycle ergometer, 60-70% heart rate reserve) hypertrophy resistance training (2sets, 10-12 repetitions, 70% of the one-repetition maximum) endurance resistance training (2 sets, 25-30 repetitions, 40% of the one-repetition maximum)
  Other Names: training intervention; resistance training

SUMMARY:
Skeletal muscle accounts for up to 40% of the total body weight and is responsible for approximately 75% of the whole body insulin-stimulated glucose uptake. Resistance training has been shown to improve insulin-stimulated glucose uptake in patients with T2DM. Therefore the investigators aim to compose the effects of 2 different resistance training protocols in combination with aerobic endurance training (AET) on muscle strength, muscle mass and glycemic control in type 2 diabetes mellitus patients (T2DM).

The investigators aim to perform an 8 week randomized controlled training intervention in 32 T2DM patients. Patients will be randomly assigned to AET (cycle ergometer, 60-70% of heart rate reserve) combined with hypertrophy resistance training (HRT, n=16, 2 sets, 10-12 repetitions, 70% of the one-repetition maximum) or with endurance resistance training (ERT, n=16, 2 sets, 25-30 repetitions, 40% of the one-repetition maximum). Body composition, blood analyses, physical work capacity and muscle strength will be measured pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus

Exclusion Criteria:

* myocardial infarction within the last 6 months
* unstable angina pectoris
* left ventricular ejection fraction less than 40%
* orthopedic limitations that eliminate to perform resistance training

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 8 weeks
  Measruement will be performed using Concept Dyno 2

SECONDARY OUTCOMES:
Muscle mass | 8 weeks
  Muscle mass will be measured using dual X-ray absorbiotometry
Glycemic control | 8 weeks
  Fasting blood glucose, HbA1c, and fructosamin will be measured using routine laboratory methods

CONTACTS AND LOCATIONS:
Overall Officials: Josef Niebauer, MD, PhD, MBA, Principal Investigator — Paracelsus Medical University
Locations (1):
- Institute of Sports Medicine, Prevention and Rehabilitation, Paracelsus Medical University, Salzburg, Austria

REFERENCES:
- [Background] Maiorana A, O'Driscoll G, Cheetham C, Dembo L, Stanton K, Goodman C, Taylor R, Green D. The effect of combined aerobic and resistance exercise training on vascular function in type 2 diabetes. J Am Coll Cardiol. 2001 Sep;38(3):860-6. doi: 10.1016/s0735-1097(01)01439-5. PMID 11527646
- [Background] Cauza E, Hanusch-Enserer U, Strasser B, Ludvik B, Metz-Schimmerl S, Pacini G, Wagner O, Georg P, Prager R, Kostner K, Dunky A, Haber P. The relative benefits of endurance and strength training on the metabolic factors and muscle function of people with type 2 diabetes mellitus. Arch Phys Med Rehabil. 2005 Aug;86(8):1527-33. doi: 10.1016/j.apmr.2005.01.007. PMID 16084803
- [Background] Castaneda F, Layne JE, Castaneda C. Skeletal muscle sodium glucose co-transporters in older adults with type 2 diabetes undergoing resistance training. Int J Med Sci. 2006;3(3):84-91. doi: 10.7150/ijms.3.84. Epub 2006 May 17. PMID 16761076
- [Background] Boule NG, Haddad E, Kenny GP, Wells GA, Sigal RJ. Effects of exercise on glycemic control and body mass in type 2 diabetes mellitus: a meta-analysis of controlled clinical trials. JAMA. 2001 Sep 12;286(10):1218-27. doi: 10.1001/jama.286.10.1218. PMID 11559268
- [Background] Dunstan DW. Aerobic exercise and resistance training for the management of type 2 diabetes mellitus. Nat Clin Pract Endocrinol Metab. 2008 May;4(5):250-1. doi: 10.1038/ncpendmet0790. Epub 2008 Mar 25. No abstract available. PMID 18364704
- [Background] Sigal RJ, Kenny GP, Boule NG, Wells GA, Prud'homme D, Fortier M, Reid RD, Tulloch H, Coyle D, Phillips P, Jennings A, Jaffey J. Effects of aerobic training, resistance training, or both on glycemic control in type 2 diabetes: a randomized trial. Ann Intern Med. 2007 Sep 18;147(6):357-69. doi: 10.7326/0003-4819-147-6-200709180-00005. PMID 17876019
- [Background] Ibanez J, Gorostiaga EM, Alonso AM, Forga L, Arguelles I, Larrion JL, Izquierdo M. Lower muscle strength gains in older men with type 2 diabetes after resistance training. J Diabetes Complications. 2008 Mar-Apr;22(2):112-8. doi: 10.1016/j.jdiacomp.2007.06.008. PMID 18280441
- [Background] Tokmakidis SP, Zois CE, Volaklis KA, Kotsa K, Touvra AM. The effects of a combined strength and aerobic exercise program on glucose control and insulin action in women with type 2 diabetes. Eur J Appl Physiol. 2004 Aug;92(4-5):437-42. doi: 10.1007/s00421-004-1174-6. PMID 15232701
- [Background] Ibanez J, Izquierdo M, Arguelles I, Forga L, Larrion JL, Garcia-Unciti M, Idoate F, Gorostiaga EM. Twice-weekly progressive resistance training decreases abdominal fat and improves insulin sensitivity in older men with type 2 diabetes. Diabetes Care. 2005 Mar;28(3):662-7. doi: 10.2337/diacare.28.3.662. PMID 15735205
- See also: Institute of Sports Medicine, Prevention and Rehabilitation, Paracelsus Medical University — http://www.salk.at/sportmedizin.html